CLINICAL TRIAL: NCT05595525
Title: A Prospective, Single-center, Double-blinded, Randomized, Split-face Study Evaluating 1064nm Versus 755nm Picosecond Lasers With Diffractive Lens Array for Improvement of Skin Quality
Brief Title: Laser Treatment to Improve Skin Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pico-Skin-Quality-2022-09
Record Dates: First submitted 2022-10-20; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Skin Quality
Keywords: wrinkles; fine lines; sun spots; laxity; facial laxity
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Intervention Model Description: subjects will be randomized to have either their right facial half or left facial half treated with the 1064nm picosecond laser with diffractive lens array. The contralateral facial half not randomized will be treated with the 755nm picosecond laser with diffractive lens array.
Who Masked: Participant, Investigator
Masking Description: the blinded investigator will complete the Scientific Assessment Scale of Skin Quality (SASSQ). , the blinded investigator will complete the Physician Global Aesthetic Improvement Scale (PGAIS) and percent improvement evaluation. Percent Improvement Evaluation by Blinded investigator .
  Subjects are blinded to which side receives which laser
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A = right side face treated with 1064nm and left with 755nm (Experimental): subject will have their right half of their face treated with the 1064nm picosecond laser with diffractive lens array. Then the contralateral, left half will be treated with the 755nm picosecond laser with diffractive lens array. Subjects will receive three (3) treatments, four (4) weeks ± 7 days apart to each facial half.
  Interventions: Device: 1064NM pico Laser; Device: 755NM pico Laser
- Group B = left side face treated with 1064nm and right with 755nm (Experimental): subject will have their left half of their face treated with the 1064nm picosecond laser with diffractive lens array. Then the contralateral, right half will be treated with the 755nm picosecond laser with diffractive lens array. Subjects will receive three (3) treatments, four (4) weeks ± 7 days apart to each facial half.
  Interventions: Device: 1064NM pico Laser; Device: 755NM pico Laser

INTERVENTIONS:
Device: 1064NM pico Laser — There have been small studies demonstrating the use of picosecond lasers for treatment of wrinkles and skin laxity; however, there have been no studies investigating the use of picosecond lasers for the overall improvement in skin quality.
  Other Names: Candela 1064NM Laser
Device: 755NM pico Laser — There have been small studies demonstrating the use of picosecond lasers for treatment of wrinkles and skin laxity; however, there have been no studies investigating the use of picosecond lasers for the overall improvement in skin quality.
  Other Names: Cynosure 755NM Laser

SUMMARY:
To assess the efficacy of a 1064nm picosecond laser (PicoWay; Candela; Marlborough, MA) with diffractive lens array and a picosecond 755nm laser (PicoSure®; Cynosure®; Westford, MA) with diffractive lens array in subjects for the improvement of facial skin quality. Secondary objectives of this clinical trial are to assess whether the 1064nm or 755nm picosecond laser is more efficacious in improving facial skin quality, safety of the procedure, comfortability of the procedure, and subject satisfaction.

DETAILED DESCRIPTION:
subject will be randomized to have either their right facial half or left facial half treated with the 1064nm picosecond laser with diffractive lens array. The contralateral facial half not randomized will be treated with the 755nm picosecond laser with diffractive lens array. Subjects will receive three (3) treatments, four (4) weeks ± 7 days apart to each facial half.

For additional comfort, cold air cooling (Zimmer MedizinSystems, Irvine, CA) set on level 5 will be used throughout the treatment. After each treatment, subjects will be provided with CeraVe gentle facial cleanser (CeraVe; New York, NY) and CeraVe lotion (CeraVe; New York, NY) to be used twice daily for two weeks. Additionally, a mineral CeraVe sunscreen (CeraVe; New York, NY) will also be provided to subjects to be used every morning with reapplication every two (2) hours if going outside for the entirety of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged 18 to 65 years
* Fitzpatrick skin types I-VI
* Subjects in good general health based on investigator's judgment and medical history
* Must be willing to give and sign an informed consent form and photographic release form
* Willingness to have facial exams and digital photographs performed of the face
* Physician evaluator classifying the subject as moderate or severe in all categories of the Scientific Assessment Scale of Skin Quality (SASSQ): elasticity, wrinkles, skin surface roughness, lentigines/pigmentation, erythema, blemishes, and pore size
* No change in topical skin care regimen for duration of study
* Must be willing to maintain usual sun exposure
* Subject agrees to avoid tanning or use of sunless tanner during the entire course of the study
* Negative urine pregnancy test result at the time of study entry (if applicable)
* For female subjects of childbearing potential, must be willing to use an acceptable form of birth control during the entire course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment.

  1. A female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation.
  2. Acceptable methods of birth control are: oral contraceptives, contraceptive patches/rings/implants, Implanon®, Depo-Provera®, double-barrier methods (e.g., condoms and spermicide), abstinence, and/or vasectomy of partner with a documented second acceptable method of birth control, should the subject become sexually active.
* Must be willing to comply with study treatments and complete the entire course of the study

Exclusion Criteria:

* Mesotherapy, dermal fillers, biostimulatory injectables, and/or fat grafting in the treatment area during the 12-month period before study treatment
* Energy-based device (i.e., radiofrequency device treatments, microfocused ultrasound device or other ultrasound-based device treatments, laser and light-based device treatments, microneedling) treatment in the treatment area in the last 6 months
* Surgery (i.e., face lift, eyebrow lift, neck lift or lower rhytidectomy, liposuction to the neck and/or submentum, etc.) during the 12-month period before study treatment
* Chemical peel or microdermabrasion of the face within 30 days prior to enrollment in the study
* Any investigational treatment for improvement of skin quality and/or photodamage of facial skin during the 12-month period before the study treatment
* Recent use of topical tretinoin, adapalene, tazarotene, hydroquinone, imiquimod, 5- fluorouracil, ingenol mebutate, concentrated hydrogen peroxide or diclofenac to the face within the previous 2 weeks
* Creams/cosmeceuticals and/or home therapies to prevent or treat photodamage, uneven skin pigmentation, excessive erythema (redness), fine lines/wrinkles, skin laxity and/or pore size during the 4-week period before study treatment
* Subjects with scarring in the treatment areas
* Subjects with tattoos or permanent implants in the treatment areas
* Subjects with a significant history or current evidence of a medical, psychological, or other disorder that, in the investigator's opinion, would preclude enrollment into the study
* Subjects with a history of or presence of any skin condition/disease (including but not limited to any visible rash, atopic dermatitis, psoriasis, actinic keratoses, keratinocyte carcinoma, melanoma, etc.) in the treatment area that might interfere with the diagnosis or evaluation of study parameters
* Skin with open wounds, excessively sensitive skin, neurotic excoriations, dermatitis or inflammatory rosacea in the treatment area
* History of keloid or hypertrophic scarring
* Subjects with an active bacterial, viral, or fungal infection of the treatment areas
* Subjects who spray tanned or used sunless tanners in the treatment areas four (4) weeks prior to study treatment
* History of lidocaine and/or tetracaine sensitivity deemed by the investigator to preclude the subject from enrolling into the study
* Individuals with known allergies or sensitivities to any of the ingredients of any topical products being used in this study
* Subjects on systemic steroids (i.e., prednisone, dexamethasone), or topical steroids on the face which should be rigorously avoided prior to and throughout the course of treatment
* Subjects planning any cosmetic procedure to the treatment areas during the study period, other than the treatment that will be performed by the investigator
* Presence of incompletely healed wound(s) in the treatment area
* Subjects who are on an immunosuppressant or have an autoimmune condition
* Female subjects who are pregnant, planning a pregnancy, or breast feeding during the study
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Scientific Assessment Scale of Skin Quality (SASSQ) to assess change | Screening, Baseline, Day 28, Day 56, Day 140
  Scientific Assessment Scale of Skin Quality (SASSQ) (circle one)
  Elasticity
  0- No 1- Mild 2- Moderate 3- Severe 4- Very Severe
  Wrinkles
  0- No 1- Mild 2- Moderate 3- Severe 4- Very Severe
  Skin Surface Roughness
  0- No 1- Mild 2- Moderate 3- Severe 4- Very Severe
  Lentigines/ Pigmentation
  0- No 1- Mild 2- Moderate 3- Severe 4- Very Severe
  Erythema
  0- No 1- Mild 2- Moderate 3- Severe 4- Very Severe
  Pore Size
  0- Fine 1- Small 2- Moderate 3- Large 4- Very Large
Physician Global Aesthetic Improvement Scale (PGAIS) by blinded investigator to assess change | Day 28, Day 56, Day 140
  Blinded Physician Global Aesthetic Improvement Scale Assessment (PGAIS) Rating Description
  1. Very Much Improved: Optimal cosmetic result in this subject.
  2. Much Improved: Marked improvement in appearance from the initial condition, but not completely optimal for this subject.
  3. Improved: Obvious improvement in appearance from initial condition, but a re- treatment is indicated.
  4. No Change: The appearance is essentially the same as the original condition.
  5. Worse: The appearance is worse than the original condition. Scores (write a number under each treated area or check "Not Treated")
  Left Facial Half Right Facial Half
  Not Treated Not Treated
Percent improvement of skin quality by blinded investigator to assess change | Day 28, Day 56, Day 140
  Blinded Investigator Percent Improvement Evaluation - Left Facial Half Degree of improvement from clinical evaluation, compare to baseline, using a 1-10 scale.
  1 (0-10%) 2 (10-20%) 3 (20-30%) 4(30-40%) 5 (40-50%)
  6 (50-60%) 7 (60-70%) 8 (70-80%) 9 (80-90%) 10 (90-100%)
  Blinded Investigator Percent Improvement Evaluation - Right Facial Half Degree of improvement from clinical evaluation, compare to baseline, using a 1-10 scale.
  1 (0-10%) 2 (10-20%) 3 (20-30%) 4(30-40%) 5 (40-50%)
  6 (50-60%) 7 (60-70%) 8 (70-80%) 9 (80-90%) 10 (90-100%)

SECONDARY OUTCOMES:
Subject Global Aesthetic Improvement Scale (SGAIS) | Day 28, Day 56, Day 140
  Subject Global Aesthetic Improvement Scale Assessment (SGAIS) How would you rate the change in appearance of your treated areas? Non-treated areas will be checked as "Not Treated" for you.
  Rating Description
  1. Very Much Improved: Optimal cosmetic result
  2. Much Improved: Marked improvement in appearance form the initial condition, but not completely optimal
  3. Improved: Obvious improvement in appearance from initial condition
  4. No Change: The appearance is essentially the same as the original condition
  5. Worse: The appearance is worse than the original condition Scores (write a number to rate each treated area)
  Left Facial Half Right Facial Half
  Not Treated Not Treated
Subject Satisfaction Questionnaire | Day 140
  Subject Satisfaction Questionnaire How would you rate your satisfaction of each treated area? Non-treated areas will be checked as "Not Treated" for you.
  Rating Description 0 Not satisfied
  1. Somewhat satisfied
  2. Satisfied
  3. Very satisfied
  4. Extremely Satisfied Scores (write a number to rate each treated area)
  Left Facial Half Right Facial Half
Comfort level visual analog scale post-procedure by subjects | Baseline, Day 28, Day 56
  Visual Analog Scale - Left Facial Half Visual Analog Scale (Circle One)
  1 2 3 4 5 6 7 8 9 10
  Visual Analog Scale - Right Facial Half Visual Analog Scale (Circle One)
  1 2 3 4 5 6 7 8 9 10
Evaluation of side effects and adverse effects by investigators | Baseline, Day 28, Day 56, Day 140
  Treating Investigator Evaluation of Side Effects Rating Description 0 NONE: Normal
  1. TRACE: Barely visible and localized
  2. MILD: Somewhat visible and diffuse
  3. MODERATE: Visible and diffuse
  4. SEVERE: Extremely visible and dense SCORES (write number under each treated area or check "Not Treated") Erythema Left Facial Half Right Facial Half
  Edema Left Facial Half Right Facial Half
  Hyperpigmentation Left Facial Half Right Facial Half
  Hypopigmentation Left Facial Half Right Facial Half
  Bruising Left Facial Half Right Facial Half
  Ulcer Left Facial Half Right Facial Half

IPD SHARING:
Plan to Share IPD: Undecided